CLINICAL TRIAL: NCT01889615
Title: Dual PETOvac - Dual Time PET/CT in the Preoperative Assessment of Ovarian Cancer
Acronym: Dual PETOvac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mie Holm Vilstrup, MD, Odense University Hospital
Other Study IDs: NMA K70 Dual PETOvac
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; PET/CT; glucose 6 phosphatase
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tissue samples from the ovarian cancer and metastasis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected ovarian cancer: dual time PET/CT
  Interventions: Other: PET/CT(3hours]

INTERVENTIONS:
Other: PET/CT(3hours] — Low dose PET/CT 1 and 3 hours after injection of FDG, followed by a diagnostic CT with iv contrast
  Other Names: Dual time PET/CT: PET 1 and 3 hours after injection of FDG

SUMMARY:
The investigators want to compare the use of MRI with PET/CT preformed after 1 hour and 3 hours in preoperative assessment of resectability.

The investigators' hypothesis is that dual time PET/CT performed at 60 and 180 minutes will increase the diagnostic accuracy of conventional PET (performed at 60 minutes) in preoperative assessment of resectability.

Further more the investigators suggest that the GLUT/G6Pase index correlates to the SUVmax. And retention index (RI, see Methods - PET protocol) is a prognostic marker in ovarian cancer.

DETAILED DESCRIPTION:
The use of PET/CT in ovarian cancer has not been well-established.

The diagnosis usually includes physical examination (incl. pelvic examination), blood test incl. CA-125 and transvaginal ultrasound. Furthermore imaging includes CT of thorax/abdomen and/or MR of pelvic. Ninety per cent of the ovarian cancers are epithelial carcinoma (EOC), which can be divided into serous (45%), mucinous (4%), endometrioid (5%), clear cell, undifferentiated and mixed types. All EOC are treated equally.

Treatment of ovarian cancer involves surgery and chemotherapy. The decision of operability is made at the multidisciplinary conference. Prognosis depends not only in the stage and histological type of the tumor but also at the end result of surgery. Residual disease after initial surgery is a strong prognostic factor for survival, with improvement on both overall and progression free survival being greatest in women with no or minimal (tumor < 1 cm) visible disease at the end surgery. Supra radical surgery is a radical procedure plus e.g. extensive peritonectomy, resection of liver metastases, splenectomy, resection of the tail of pancreas and bowel resection. Only 60% of patients in advanced stage ovarian cancer are deemed optimal debulked peroperative. Patients with optimal debulking have a 5 year survival of 42% versus patients not possible of achieve radical operation with 5 year survival of 15%, resulting in a hazard rate of 2,12 for optimal vs. not optimal debulking. A correct preoperative assessment is important in planning of operation and to avoid futile operation in patients not resectable.

Preoperative CT has shown to have a predictive value in assessment of the completeness of cytoreduction. But also PET/CT is has shown to be a independent predictor of resectability. Currently MR is standard in evaluating patient operability.

Studies has shown PET/CT to be particularly useful in distinguishing patients with stages I-IIIB and IIIC-IV, with an accuracy of 98% compared to 88% with CT alone. The latter group is important to identify because optimal debulking often is not possible and they will benefit from preoperative chemotherapy. Currently the use of PET/CT in staging ovarian cancer is controversial, mainly because of the relatively low specificity, due to FDG-uptake in inflammatory cells and benign lesions. The concordance of PET/CT and surgical staging of ovarian cancer have been reported to range from 69% to 78%.8,9, And a recent study found good correlation between PET/CT findings and laparoscopy but a high rate of false negative results in lesions < 5 mm. But dual time point imaging is maybe the solution to this problem. Today it is standard to perform PET/CT scan 60-90 minutes after injection of tracer. Theoretically, you should get increased tumor/background ratio by performing a late scan, thus better being able to distinguish between malignant and benign. Dual time imaging studies in head and neck cancers, breast cancer and lung cancer suggests improvement in diagnostic accuracy of PET. But the use of delayed imaging in ovarian cancer has not been studied.

The tracer used in PET is 18F-fluoro-2-deoxy-d-glucose. Generally cancer cells are thought to have low or absent G6Pase expression compared to normal cells and cancer cells have increased expression of GLUT (especially GLUT1) and hexokinase (especially HK2), which further leads to intracellular trapping of FDG-6-phosphate in malignant cells and there by yielding high maximum standardized uptake value (SUVmax). But ovarian cancers have found to have a relatively low ratio of hexokinase/phosphatase maybe explaining the low/absent rise in FDG-uptake. The amounts of GLUT, hexokinase and G6Pase are responsible for the FDG trapping intracellular and the retention on the late scans.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of ovarian cancer
* Referred to Department of Gynecology, OUH

Exclusion Criteria:

* Unable to corporate to MR
* Diabetes Mellitus
* Prescan glucose level > 10 mmol/l (PET)
* non-ovarian cancer (incl. benign)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy in MR, PET/CT 1h and 3h preoperative assessment of ovarian cancer resectability(PET/CT[1]) of the radioactive tracer FDG with PET/CT performed after 3 hours (PET/CT[3]) in a group of patients with high suspicion of ovarian cancer | 2 years
  At biweekly multidisciplinary meetings patient resectability is assessed based on disease spread by using conventional PET/CT and MR. The MR, PET [1 hour] vs. PET [3 hours] in assessment of disease spread compared to peroperative findings.

SECONDARY OUTCOMES:
Compare SUVmax with the expression of GLUT1, hexokinase and G6Pase in tumors | Immediately after surgery
  Compare the SUVmax measured on PET[1hour] and PET[3hours]with the measured expression of GLUT1, hexokinase II and G6Pase in primary tumors and metastasis

OTHER OUTCOMES:
Compare SUVmax, RI, tumor/liver ratio and GLUT1/G6Pase as a prognostic marker | 5 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mie H Vilstrup, MD, Principal Investigator — Department of Nuclear Medicine, Odense University Hospital
Locations (1):
- Department of Nuclear Medicine, Odense C, Fünen, Denmark